CLINICAL TRIAL: NCT01567930
Title: A Phase II Study of Temsirolimus as Second-line Therapy in Patients With Advanced, Unresectable Hepatocellular Carcinoma
Brief Title: Temsirolimus as Second-line Therapy in HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee Cancer Institute (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-2247
Record Dates: First submitted 2012-02-01; First posted 2012-03-30 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-03

CONDITIONS: Unresectable or Metastatic Hepatocellular Carcinoma
Keywords: Temsirolimus; HCC; Advanced hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Temsirolimus — Intervention: Temsirolimus IV Eligible patients will receive temsirolimus IV on days 1,8,15 every 21 days. Treatment will continue till disease progression or untolerable side effects
  Other Names: Torisel

SUMMARY:
The purpose of this study is to evaluate the activity of temsirolimus in patients who have advanced hepatocellular carcinoma (HCC) and have been treated with one previous chemotherapy or biologic therapy like sorafenib, but have experienced disease progression or intolerance to that therapy.

DETAILED DESCRIPTION:
Currently, no standard therapy exists for patients who progress on sorafenib. mTOR signaling is often up-regulated in HCC promoting cell growth and survival. This process is inhibited by rapamycin, a specific inhibitor of mTOR. Temsirolimus, a rapamycin analog, may delay tumor progression by inhibiting mTOR in HCC.Intervention: Temsirolimus IV

Eligible patients will receive temsirolimus IV on days 1,8,15 every 21 days. Treatment will continue till disease progression or untolerable side effects

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have advanced unresectable or metastatic hepatocellular carcinoma (HCC). Prior diagnosis of HCC could have been established histologically or based on one of the following criteria:

   * Liver mass > 2cm: Characteristic enhancement on at least one imaging technique(triphasic CT scan, MRI, or contrast enhanced ultrasound) or AFP > 200 ng/ml.
   * Liver mass between 1 and 2 cm: Characteristic enhancement on two imaging techniques.Diagnosis of HCC must have been confirmed by biopsy if non-characteristic enhancement on imaging.
2. All patients must have received exactly one prior systemic therapy (cytotoxic chemotherapy or targeted therapies) and must not be eligible for further locoregional treatment modalities.
3. All patients must have measurable disease per RECIST criteria.
4. Patients with previous locoregional therapies, including but not limited to radio-frequency ablation, cryoablation, percutaneous ethanol injection, chemo-embolization, hepatic artery embolization, and hepatic artery infused FUDR, stereotactic radiotherapy are eligible provided they have documented progression of their disease or have measurable extrahepatic disease.
5. Patients must have an ECOG performance status of 0 - 2 (see Appendix B).
6. Patients must be greater than or equal to 18 years of age.
7. Patients with Child-Pugh class A (score of 5-6) or class B (score of 7-9) are eligible.
8. Patients must have adequate organ function as defined by:

   * AST, ALT and Alkaline phosphatase ≤ 5x upper limit of normal (ULN)
   * Total Bilirubin < 2 mg/dl.
   * Creatinine clearance ≥ 15ml/min & patients must not be dialysis dependent.
9. Patients must have adequate bone marrow function as defined by:

   * Leukocytes ≥ 2000 / mm3 or absolute neutrophil count (ANC) ≥ 1000 / mm3
   * Platelet count ≥ 75000 / mm3
10. Pregnant and nursing women will be excluded from this study. All patients of reproductive potential must agree to use adequate birth control measures to be eligible for study enrollment.
11. Prior palliative radiotherapy is permissible provided it has been completed at least 2 weeks prior to study entry and the patient has recovered from any radiation-related side effects.
12. Patients must not be receiving any other investigational agents or other anti-cancer therapies. At least 28 days must have elapsed since completion of previous systemic therapy prior to study entry and the patient should have recovered from all toxicities related to prior therapy.
13. Patients must not have a history of other malignancies that are active and require therapy (other than non-melanoma skin cancers).

Exclusion Criteria:

1. Patients with prior treatment with any mTOR inhibitor are not eligible.
2. Patients with a history of an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris,cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are not eligible.
3. Patients taking cytochrome P450 enzyme-inducers or inhibitors are not eligible.
4. Patients with a known history of HIV infection are not eligible.
5. Patients with uncontrolled hyperlipidemia or hypercholesterolemia are not eligible (fasting serum cholesterol > 350 mg/dL or fasting serum triglycerides > 400 mg/dL).
6. Patients with a known history or clinical evidence of CNS metastases are not eligible.
7. Patients who, in the best judgment of the investigator, will not be able to comply with the requirements of the protocol are not eligible.
8. Patients with Child-Pugh class C liver disease are not eligible.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Disease Progression
  The primary outcome measure is to determine the proportion of patients who are progression free at 3 months.

SECONDARY OUTCOMES:
Response rate
  Response rate, clinical benefit rate (complete + partial response + stable disease > 12 weeks) and overall survival with temsirolimus
Safety and tolerability
  Number and frequency of adverse events and serious adverse events will be monitored.
Biochemical response
  Biochemical response (>50% decline in AFP levels from baseline) with temsirolimus
Pharmacokinetics
  Pharmacokinetics will be assessed: AUC pre-dose, 1, 3, 24,48, 72 and 162 hours post dose.
Circulating tumor cells levels
  Feasibility and utility of circulating tumor cells in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Jasgit Sachdev, MD, Principal Investigator — University of Tennessee Cancer Institute
Locations (1):
- Boston Baskin Cancer Foundation, Memphis, Tennessee, United States